CLINICAL TRIAL: NCT03802292
Title: First-In-Man, Phase I, Single-Blind, Placebo-Controlled, Ascending Single Dose Study of Intravenous YQ23 in Healthy Male and Female Subjects to Assess Safety, Tolerability, and Pharmacokinetics
Brief Title: First-In-Man, Healthy Volunteer Study to Evaluate Safety on the Use of YQ23
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Beta Innovation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: NBI(CT)-YQ23-2015-001
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Dose escalation study to determine the safe dose level.
Who Masked: Participant
Masking Description: Single blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose YQ23 (Active Comparator)
  Interventions: Biological: YQ23
- Single Dose Placebo (Placebo Comparator)
  Interventions: Biological: Matching Placebo

INTERVENTIONS:
Biological: YQ23 — Single dose of YQ23 delivered via intravenous route. Ascending dose levels will be evaluated
  Arms: Single Ascending Dose YQ23
Biological: Matching Placebo — Single dose of the matching placebo delivered via intravenous route.
  Arms: Single Dose Placebo

SUMMARY:
This study is to test the safety, tolerability, pharmacokinetics (PK-the amount of study drug in the blood), and immunogenicity (how the study drug affects the immune system) of single dose and dose levels of an investigational drug called YQ23.

DETAILED DESCRIPTION:
This is a first-in-man, phase 1, single-blind, randomized, placebo-controlled study in healthy volunteers. It will be conducted at a single centre and will enroll approximately 64 subjects. Subjects will either receive a single dose of study drug or placebo in a 3:1 ratio. Eight dose levels of YQ23 will be evaluated.

Each dose level group will be divided into 2 cohorts, with each cohort being dosed at last 24 hours apart. The leading cohort will comprise of 2 subjects, with 1 subject receiving YQ23 and 1 subject receiving placebo. The remaining cohort will comprise of 6 subjects, with 5 receiving YQ23 and 1 receiving placebo.

Safety assessments will be performed throughout the dosing and follow-up periods, and multiple PK samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any ethnic origin, between 18 and 50 years of age, inclusive.
* Body mass index between 18.0 and 30.0 kg/m2, inclusive, and body weight between 50 and 100 kg, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations (congenital non-hemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check in, as assessed by the Investigator (or designee).
* Females of non-childbearing potential defined as permanently sterile (ie, due to hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or postmenopausal (defined as at least 12 months postcessation of menses without an alternative medical cause and follicle stimulating hormone level ≥ 40 mIU/mL). Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception as detailed in the protocol.
* Able to comprehend and willing to sign an Informed Consent Form and to abide by the study restrictions.
* Subjects must agree to receive a bovine product.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance (excluding non-active hay fever), unless approved by the Investigator (or designee).
* Any abnormality in the 12-lead ECG that, in the opinion of the Investigator (or designee), increases the risk of participating in the study.
* Any clinically relevant findings on echocardiography, including left ventricular ejection fraction < 50% at baseline.
* Supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 bpm, respectively, or lower than 90/50 mmHg and 40 bpm, respectively, at Screening or Check-in, confirmed by a repeat measurement.
* Liver function test results for aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), and/or bilirubin > 1.5 x Upper Limit of Normal (ULN) at Screening or Check-in confirmed by repeat measurement.
* Total red blood cell count, total white blood cell count, and/or haemoglobin levels outside of the normal reference range at Screening or Check-in, confirmed by repeat measurement.
* History of alcoholism or drug/chemical abuse within 2 years prior to Check in.
* Alcohol consumption of > 21 units per week for males and > 14 units for females.
* Positive alcohol breath test result or positive urine drug screen (confirmed by repeat) at Screening or Check in.
* Positive hepatitis panel and/or positive human immunodeficiency virus test.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
* Use or intend to use any prescription medications/products other than hormone replacement therapy (HRT), oral, implantable, transdermal, injectable, or intrauterine contraceptives within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use slow release medications/products considered to still be active within 14 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
* Use or intend to use any non-prescription medications/products (with the exception of vitamins/mineral supplements) and phytotherapeutic/herbal/plant derived preparations within 7 days prior to dosing, unless deemed acceptable by the Investigator (or designee).
* Smoke more than 10 cigarettes or use the equivalent tobacco or nicotine containing products per day.
* Receipt of blood products within 2 months prior to Check in.
* Receipt of bovine Haemoglobin-based Oxygen Carrier (HBOC) or other HBOC in the past.
* Donation of blood from 3 months prior to Screening, plasma from 7 days prior to Screening, or platelets from 6 weeks prior to Screening, or donations on more than 2 occasions within the 12 months preceding dosing.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study.
* Have known allergies to bovine products.
* Are vegetarians.
* Subjects who have had a clinically significant illness as determined by the Investigator within 4 weeks of the start of dose administration.
* Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the incidence of Treatment-emergent Adverse Events (TEAE) | From the time of signing the Informed Consent Form to final discharge from the study (approximately 8 weeks)
  Number of TEAEs will be listed according to the severity (mild, moderate, severe) as assessed by the Investigator.
Safety as assessed by the incidence of laboratory abnormalities, based on haematology, clinical chemistry, and urinalysis test results | From the time of signing the Informed Consent Form to D8 visit (approximately 36 days)
  All serum biochemistry, haematology, and urinalysis data outside the clinical reference ranges will be listed by parameter and treatment.
Safety as assessed by 12-lead electrocardiogram (ECG) | From the time of signing the Informed Consent Form to D8 visit (approximately 36 days)
  ECG parameters such as PR, QRS, QT and QTcF in milliseconds will be recorded. Clinically significant abdominal findings will be reported as Adverse Events (AE).
Safety as assessed by echocardiogram | From the time of signing the Informed Consent Form to D2 visit (approximately 30 days)
  Clinically significant abnormal echocardiogram findings will be recorded as AEs.
Safety as assessed by vital sign measurement of blood pressure | From From the time of signing the Informed Consent Form to D8 visit (approximately 36 days)
  Systolic and Diastolic blood pressure (in mmHg) which is outside the clinical reference ranges and considered as clinically significant will be reported as AE.
Safety as assessed by vital sign measurement of pulse rate | From From the time of signing the Informed Consent Form to D8 visit (approximately 36 days)
  Pulse rate (in beats/min) which is outside the clinical reference ranges and considered as clinically significant will be reported as AE.
Safety as assessed by vital sign measurement of oral body temperature | From From the time of signing the Informed Consent Form to D8 visit (approximately 36 days)
  Body temperature (in degree Celsius) which is outside the clinical reference ranges and considered as clinically significant will be reported as AE.
Safety as assessed by local tolerability assessment: pain | From the time before dosing to D3 post dose (3 days)
  The intravenous (IV) infusion site will be assessed for pain according to the following scale [Grade 0=none, 1=does not interfere with activity, 2=interferes with activity or requires repeated use of non-narcotic pain medication, 3=prevent daily activity or requires repeated use of narcotic pain medication, 4=requires medical intervention greater than analgesia]. Grade 3 or above will be recorded as AE.
Safety as assessed by local tolerability assessment: edema | From the time before dosing to D3 post dose (3 days)
  The intravenous (IV) infusion site will be assessed for edema according to the following scale [Grade 0=0 to 24mm, 1=25 to 50mm and not interfere with activity, 2=51 to 100mm, or interferes with activity, 3=more than 100mm, and interferes with daily activity, 4=necrosis]. Grade 3 or above will be recorded as AE.
Safety as assessed by local tolerability assessment: erythema intensity | From the time before dosing to D3 post dose (3 days)
  The intravenous (IV) infusion site will be assessed for erythema intensity according to the following scale [Grade 0=None, 1=light pink, 2=pinkish red, 3=intense red]. Grade 3 or above will be recorded as AE.
Safety as assessed by local tolerability assessment: erythema size | From the time before dosing to D3 post dose (3 days)
  The intravenous (IV) infusion site will be assessed for erythema size according to the following scale [Grade 0=0 to 24mm, 1=25 to 50mm, 2=51 to 100mm, 3=more than 100mm, 4=necrosis or exfoliative dermatitis]. Grade 3 or above will be recorded as AE.

SECONDARY OUTCOMES:
Pharmacokinetics of YQ23 as assessed by Area under curve (AUC) on all subjects | From study Day 1 (dosing of study drug) until Day 4 of trial participation.
  Plasma levels of YQ23 will be serially evaluated following dosing of study drug, and the AUC will be calculated.
Pharmacokinetics of YQ23 as assessed by the maximum concentration of YQ23 on all subjects | From study Day 1 (dosing of study drug) until Day 4 of trial participation.
  Plasma levels of YQ23 will be serially evaluated following dosing of study drug, and the maximum plasma concentration (Cmax) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Billy Lau, PhD, Study Director — New Beta Innovation Limited
Locations (1):
- Covance CRU Limited, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No